CLINICAL TRIAL: NCT06433583
Title: Pilot Study on the Acceptability of Auricular Vagus Nerve Neurostimulation for the Prevention of Non-suicidal Self-injury Recurrence in Adolescents
Brief Title: Pilot Study on the Acceptability of Auricular Vagus Nerve Neurostimulation in Adolescents
Acronym: NEUROMUTE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Régional Metz-Thionville (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2023-01-CHRMT
Record Dates: First submitted 2024-05-23; First posted 2024-05-29 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Psychiatric Disorder
Keywords: non-suicidal self-injury; transcutaneous auricular vagal nerve stimulation
MeSH Terms: conditions — Mental Disorders; Self-Injurious Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- transcutaneous auricular vagal nerve stimulation (taVNS) treatment (Experimental)
  Interventions: Device: transcutaneous auricular vagal nerve stimulation

INTERVENTIONS:
Device: transcutaneous auricular vagal nerve stimulation — The use of TENS ECO PLUS and the vagus nerve ear electrode medical devices for transcutaneous auricular vagal nerve stimulation (taVNS) everyday for 10 minutes twice a day or 20 minutes for 8 successive weeks. Patients are included at week 0, use taVNS between week 2 and 10, and are followed up until week 22.
  Patient adherence: percentage of patients performing 20 minutes of daily stimulation on at least 5 days a week for at least 6 cumulative weeks.

SUMMARY:
Non-suicidal self-injury (NSSI) are acts defined by the DSM-5 (Diagnostic and Statistical Manual of Mental Disorders 5) as intentional and deliberate, occurring outside a psychotic state and directly causing moderate injury.

Their international prevalence is between 13 and 17% in adolescents and young adults, and has recently increased with the COVID-19 health crisis, with the prevalence of NSSI rising to 40% in adolescents. Access to psychiatrists is declining. Drug solutions, meanwhile, lack scientific proof in this indication.

The autonomic nervous system and the hypothalamo-hypophyseal axis are involved in the human response to experimentally-induced pain, as well as in stress regulation, notably via control of cortisol secretion.

Abnormally low levels of the latter hormone have been detected in persons with NSSI disorder.

Transcutaneous neurostimulation of the atrial vagus nerve (taVNS) has been studied for some ten years. The afferent branches of the vagus nerve stimulate the hypothalamic-pituitary axis, leading to the production of cortisol by the adrenals.

The hypothesis of this research is that stimulation of the vagus nerve by taVNS would improve the functioning of the hypothalamic-pituitary axis in patients with NSSI, and thus reduce the frequency of acting out.

Although taVNS is an easy-to-access technique that patients can implement at home, the question of adherence to this treatment in adolescents has not yet been evaluated. The aim of this pilot study is to assess whether adolescents with NSSI will adhere to taVNS treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents aged between 13 and 17 years old
* Patients with NSSI disorder as defined by DSM-5
* Patient affiliated to a social security scheme
* Patient who parents or guardians have signed a free and informed consent form
* Patient able to understand neurostimulation instructions

Exclusion Criteria:

* Contraindication to taVNS:
* Malformation, skin pathology of the external ear. (piercings in the area concerned must be removed during the neurostimulation session).
* Children with sleep apnea syndrome treated with NIV (non-invasive ventilation)
* Presence of epileptic seizures
* Proven cardiac pathology on the advice of the attending cardiologist
* History of venous or arterial thrombosis
* Adolescent with pacemaker or defibrillator
* Adolescent with an active implantable device
* Pregnancy (based on anamnestic criteria, checked by blood test if necessary)
* Patients with psychotic episodes, confusional states or severe neurodevelopmental disorders
* Patients with an allergic skin reaction to silicone (component of the ear electrode)
* Patients with a cochlear implant on the stimulation side
* Pregnant or breast-feeding women
* Minor under guardianship
* Minor under judicial measure or sanction

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 22 (Estimated)
Dates: Start 2024-11-28 (Actual); Primary Completion 2027-05-28 (Estimated); Study Completion 2027-05-28 (Estimated)

PRIMARY OUTCOMES:
Patient adherence to treatment | 10 weeks after inclusion
  percentage of patients performing 20 minutes of daily stimulation on at least 5 days a week for at least 6 weeks.

SECONDARY OUTCOMES:
Other caracteristics for patient adherence to treatment | 10 weeks after inclusion
  Cumulative daily duration of stimulation, number of daily taVNS sessions performed, number of days per week with at least one session, number of weeks with at least one session, number of premature study exists and reasons.
Frequency of weekly non-suicidal self-injury (NSSI) | weekly, from 2 weeks before treatment and up to 20 weeks after treatment
  Assessed by the patient on a Likert scale in a logbook.
Anxiety and depression levels | at week 0, 2, 10 and 22 after inclusion
  Using the Hospital Anxiety Depression (HAD) scale The Hospital Anxiety and Depression Scale (HADS) is a 14-item measure designed to assess anxiety and depression symptoms in medical patients, with emphasis on reducing the impact of physical illness on the total score.
  Items are rated on a 4-point severity scale. The HADS produces two scales, one for anxiety (HADS-A) and one for depression (HADS-D), differentiating the two states. Scores of greater than or equal to 11 on either scale indicate a definitive case.
Adverse events | up to 22 weeks after inclusion
  assessed through patient logbook and consultations with psychiatrist during taVNS treatment
Patient's experience of taVNS | at week 10 after inclusion
  Semi-structured questionnaire at the end of taVNS.

CONTACTS AND LOCATIONS:
Overall Officials: Dorin SINDILA, MD, Principal Investigator — CHR Metz Thionville
Locations (1):
- Centre Médico-Psychologique adolescents - CHR Metz-Thionville, Thionville, France

IPD SHARING:
Plan to Share IPD: No